CLINICAL TRIAL: NCT01144988
Title: An Academic Prospective Single-arm Phase II Clinical Trial for Evaluation of Advanced Functional Neuroimaging Techniques and Molecular Markers in the Course of Anti-angiogenic Therapies in Malignant Gliomas
Brief Title: Avastin / Irinotecan in Patients With Recurrent or Progressive Malignant Glioma
Acronym: AVIRMA01-09
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Roche, Austria (Unknown)
Responsible Party: Stockhammer, Guenther, MD, Prof., Medical University Innsbruck, Department for Neurology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EUDRACT-Nr: 2009-015036-15
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Recurrent Malignant Glioma
Keywords: Recurrent Malignant Glioma; Bevacizumab / Irinotecan; Functional MR Imaging; Metabolic Imaging (FET/FLT-PET)
MeSH Terms: conditions — Glioma | interventions — Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab / Irinotecan — Bevacizumab (10mg/kg KG) Irinotecan (125 mg/ m2 or 340 mg/m2 depending on usage of EIAED)

SUMMARY:
Malignant glioma are the most common and aggressive primary brain tumors in adults. Despite advances in multimodal treatment including surgery, radiation and chemotherapy, most patients have a dismal prognosis of 9-15 months (Stupp et al., NEJM 2005).

A major reason for the aggressiveness of malignant glioma is a pronounced tumor neovascularization, mainly driven by the vascular endothelial growth factor (VEGF) and its receptors. The therapeutic monoclonal antibody Bevacizumab (Avastin®) inhibits the VEGF pathway by binding the VEGF ligand. In Magnetic Resonance Imaging (MRI) this treatment reduces contrast enhancement by restoring both, the blood-brain-barrier and the destabilized vessel integrity. Furthermore, it raises the sensitivity of co-administered chemotherapeutics such as Irinotecan. In conclusion, anti-angiogenic therapy leads to the problem that the routinely used MRI techniques cannot distinguish anti-vascular effects from true anti-tumor effects.

The study hypothesis of the clinical trial part is that in 35% of malignant glioma patients Avastin / Irinotecan chemotherapy results in objective tumor responses assessed by standard / functional MRI and FET- /FLT-PET neuroimaging. The study hypothesis for the translational study part is that the expression of the molecular targets of Avastin and Irinotecan in malignant glioma tissue ( = tumor and vascular cells) are predictive for Avastin / Irinotecan therapy induced treatment response measured by functional MRI and FET- / FLT-PET imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients present with a first or second tumor recurrence / progression of a histological confirmed supratentorial malignant glioma WHO Grade III-IV (Classification following WHO criteria).
2. Patients with surgical resection of tumor recurrence / progression: Following standard therapy(first recurrence) or standard therapy / second line chemotherapy (second recurrence, excepting antiangiogenic approaches) patients must have evidence of further tumor progression measured by standard MRI sequences (MacDonald criteria). If possible, patients may have prior surgical resection of the tumor progression and will be eligible if the following conditions apply:

   * Patients must have recovered from the effects of surgery
   * To adequately asses the malignant glioma before surgery and the extent of residual disease postoperatively, two MRIs scans have to be performed:
   * A first standard MRI scan has to be done within 1 week before surgery to document a progressed or recurrent malignant glioma.
   * A second standard / functional MRI scan has to be done between 24 and 48 hours after surgery to document the postoperative malignant glioma (Baseline MRI scan).
   * FET- / FLT-PET scans have to be done within 2 weeks after surgery to document the postoperative malignant glioma (Baseline PET scans).

   Patients without surgical resection of the tumor recurrence / progression: Patients must have evidence of tumor progression measured by standard MRI sequences (MacDonald criteria).
   * Additional functional MRI sequences have to be done within 1 week prior to study enrollment.
   * FET- / FLT-PET scans have to be done within 2 weeks after surgery to document the postoperative malignant glioma (Baseline PET scans).
3. Resolution of all acute toxic effects of prior therapy to grade ≤ 1 (except alopecia)
4. Patients must have an ECOG performance status of 0-2
5. Patients must be ≥ 18 years and ≤ 80 years of age, with a life expectancy of greater than 8 weeks
6. Patients must have adequate organ function as defined by the following criteria:

   Bone Marrow Reserve
   * Platelets ≥ 75.000/μL
   * Absolute Neutrophil Count ≥ 1500/μL
   * Hemoglobin ≥ 10.0 g/dL Blood Coagulation
   * aPTT ≤ 1.5 times upper limit of normal (ULN) Hepatic Function
   * ASAT and ALAT ≤ 2.5 times ULN
   * ALP ≤ 2.5 times ULN
   * Total SERUM Bilirubin < 1.5 times ULN Renal Function
   * SERUM Creatinine ≤ 1.5 times ULN Metabolism
   * SERUM Albumin ≥ 3.0 g/dL All tests must be performed ≤ 3 days prior to study enrollment. Eligibility for hemoglobin count may be reached by transfusion.
7. Signed and dated informed consent document by the patient, indicating that the patient has been informed of all the pertinent aspects of the trial prior to study enrollment.
8. Willingness and ability of the patient to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

   Exclusion Criteria:
9. The patient is active participant in another clinical trial, which investigates substances with antiangiogenic effectiveness
10. Exclusion of patients in the event of

    * surgery of a recurrent / progressed malignant glioma within 2 weeks prior to study enrollment
    * chemotherapy (Standard therapy o Second Line Chemotherapy) within 2 weeks prior to study enrollment
    * radiation therapy (Standard therapy) within4 weeks to study enrollment
    * evidence in baseline MRI of intratumoral or peritumoral hemorrhage deemed clinically significant by the treating physician (area of hemorrhage > 25% of tumor area)
11. Significant Co-Morbidities within 12 months prior to study enrollment

    * myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure
    * cerebrovascular accident including transient ischemic attack
12. Significant Co-Morbidities at Baseline Evaluation

    * Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy)
    * Pulmonary embolism within 4 weeks before study enrollment
    * A known HIV (human immunodeficiency virus) or Hepatitis B/C infection or severe acute infection
13. Anticoagulation: Current treatment with therapeutic doses of Marcoumar / Sintrom excluding thrombosis prophylaxis with low dose Heparin
14. Pregnancy, Breastfeeding and Non-Contraception

    * Female patients who are pregnant or nursing
    * Patients who are sexually active and unwilling or unable to use a medically acceptable method of contraception during the trial
15. Evidence of increased intracranial pressure

    * midline shift > 5 mm
    * headache, distinct nausea and vomiting
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart excess risk associated with study participation or study drug administration, or which would make the patient inappropriate for entry into this study. The decision to enroll the patient in this study is in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
To determine the objective tumor response criteria (RR, ORR, ORD) assessed by Standard MRI and FET-/FLT-PET during Avastin / Irinotecan chemotherapy. | three years

SECONDARY OUTCOMES:
Evaluation of the predictive / prognostic value of the VEGF pathway and tumor cell proliferation rate in tumor and vascular cells of malignant gliomas treated with Avastin / Irinotecan Chemotherapy | three years

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Stockhammer, MD, Prof., Principal Investigator — Department for Neurology, Medical University Innsbruck
Locations (2):
- Austria (2):
  - Paracelsus Medical University, Christian Doppler Klinik, Salzburg, Austria
  - Medical University Innsbruck, Department for Neurology, Innsbruck

REFERENCES:
- See also: homepage Medical University Innsbruck — http://www.i-med.ac.at